CLINICAL TRIAL: NCT06476340
Title: Outcomes of Zygomatic Fractures: Cross- Sectional Study
Acronym: ZY-PROM
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Antoinette V. J. Rozeboom, Dr., Erasmus Medical Center
Other Study IDs: ErasmusMC_2
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Zygoma Fracture
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — None, questionnaires/CBCT/3D photography/physical examination

SUMMARY:
Rationale: Facial trauma is a significant event for patients, often resulting in physical and psychological consequences. Fractures in the zygomatic bone area are common due to its unique shape and positioning in the face, disrupting facial symmetry and impacting aesthetics, functionality, and psychological well-being. The zygomatic bone, crucial for facial contour and support, is associated with complications such as diplopia, sensory disturbances, and mastication problems when fractured. Treatment aims to restore function, aesthetics, and prevent long-term deformities. Despite surgical and imaging advancements, postoperative complications like residual deformity and dissatisfaction persist. Even with achieved bone symmetry, patients may perceive asymmetry. Current literature emphasizes the need for future symmetry analyses to include both soft and hard tissues.

Objective: This study aims to evaluate the long-term outcomes of zygomatic fracture treatments at Erasmus MC from 2008 to 2023.

Study design: Cross-sectional study Study population: The study population consists of adult patients aged 18 years and above diagnosed with zygomatic fractures and treated at Erasmus MC Rotterdam between 2008 and 2023.

Intervention: Not applicable Main study parameters/endpoints: The primary endpoint is patient satisfaction and quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Cone Beam Computed Tomography (CBCT) is an advanced imaging modality utilized for high-resolution three-dimensional (3D) visualization of the maxillofacial region. It employs a rotating C-arm apparatus to project a cone-shaped X-ray beam through the patient's head, yielding detailed images with minimal distortion. CBCT is pivotal in the diagnosis and assessment of maxillofacial conditions, including zygomatic fractures, while ensuring low radiation exposure. Over the past two decades, CBCT has been extensively integrated into dental and maxillofacial imaging, with numerous studies substantiating its efficacy and safety in clinical contexts. It serves as a cornerstone in orthodontic, implantological, and trauma evaluation, supported by a substantial body of evidence validating its ability to delineate bone structures and identify fractures. Human exposure to CBCT has demonstrated a robust safety profile, characterized by radiation doses lower than those of conventional CT scans, thus imparting negligible additional risk.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   Facial trauma represents a significant event in a patient's life, often resulting in physical deformities and potential psychological consequences (1, 2). In facial trauma cases, fractures occurring in the zygomatic bone area are prevalent due to the distinctive shape and positioning within the face (3, 4). These fractures can disrupt the facial symmetry, which plays a role in the perceived aesthetics and functionality of the human face, impacting not only physical appearance but also psychological well-being and social interactions (5).

   The zygomatic bone, a critical component of the midfacial skeleton, contributes to the contour and width of the face, supports the orbit and has a functional role as the origin of one of the masticatory muscles, the masseter muscle (6). Therefore, fractures in this region can lead to a variety of complications including diplopia, enophthalmos, sensory disturbances and mastication problems (7). Treatment aims not only to restore function and aesthetics but also to prevent long-term deformities.

   Despite advancements in surgical techniques and imaging modalities (8), postoperative complications such as residual deformity, asymmetry of hard and soft tissue, and dissatisfaction with facial appearance remain remain concerns that warrant further investigation. Even when bone symmetry is achieved, patients may still report perceived asymmetry (9). Current literature, primarily focused on hard tissue symmetry, indicates the necessity of including both soft and hard tissues in future symmetry analyses (10).

   This study aims to create a detailed database of patients treated for zygomatic fractures at Erasmus MC from 2008 to June 2023. By leveraging data from electronic patient records, we intend to gather extensive demographic, clinical, and treatment-related information. Following this, patients will be invited to undergo additional evaluations including Cone Beam Computed Tomography (CBCT) scans, which offer precise imaging to assess for any residual displacement and asymmetry. For soft tissue, 3D facial photography will be used to objectively measure facial asymmetry, offering a comprehensive view of both functional and aesthetic results post-recovery. Patient satisfaction and quality of life post-treatment will be assessed through validated questionnaires (FACE-Q), providing insights into the psychological and social impacts of these injuries. Functional tests will be conducted to evaluate ocular motility and cutaneous sensory function.

   Through this multifaceted approach, the study aims to identify factors contributing to optimal outcomes and those that may predispose patients to poorer prognoses. The findings will not only enhance understanding of zygomatic fractures but also inform future clinical practices, ensuring improved patient care and satisfaction through better expectation management.
2. OBJECTIVES

Primary Objective:

The primary objective of this study is to evaluate the long-term outcomes of patients treated for zygomatic fractures at Erasmus MC from 2008 to 2023. Specifically, to assess patient satisfaction with facial appearance and overall quality of life post-treatment using validated questionnaires. This will provide insights into the psychological and social impacts of zygomatic fractures and their treatment.

Secondary Objective(s):

* Residual displacement and asymmetry A secondary objective is to assess the degree of residual displacement and asymmetry in both hard and soft tissues using Cone Beam Computed Tomography (CBCT) scans and 3D facial photography. This evaluation will determine the effectiveness of current surgical techniques in restoring facial symmetry and function.
* Functional Outcomes:

To evaluate the functional outcomes of the surgical treatment, including ocular motility, range of motion/mouthopening, cutaneous sensory function. These tests will help determine the success of the treatment in restoring normal facial function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sustained a zygomatic fracture and were treated at Erasmus MC from January 2008 to June 2023.
2. Patients aged 18 years and older at the time of the initial treatment.

Exclusion Criteria:

1. Patients with incomplete or missing electronic medical records that lack essential demographic, clinical, or treatment-related information.
2. Subsequent facial trauma: Patients who experienced additional facial trauma after the initial zygomatic fracture, which could affect the outcomes and complicate the assessment of the initial treatment.
3. Zygoma arch fracture: Patients who have a zygomatic arch fracture. This will nog influence the asymmetry or physical appearance.
4. Psychiatric or cognitive disorders: Patients with psychiatric or cognitive disorders that impair their ability to provide informed consent or complete the necessary fol-low-up evaluations and questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and above diagnosed with zygomatic fractures and treated at Erasmus MC Rotterdam between 2008 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
PROM face Q | 1 year
  The primary objective of this study is to evaluate the long-term outcomes of patients treated for zygomatic fractures at Erasmus MC from 2008 to 2023. Specifically, to assess patient satisfaction with facial appearance and overall quality of life post-treatment using validated questionnaires. This will provide insights into the psychological and social impacts of zygomatic fractures and their treatment.

IPD SHARING:
Plan to Share IPD: No